CLINICAL TRIAL: NCT04444362
Title: Protective Effect of Probacine Against Negative Gut Metabolism and Organ Dysfunction After Cardiovascular Surgery: A Randomized Controlled Trial
Brief Title: Protective Effect of Probacine Against Negative Gut Metabolism and Organ Dysfunction After Cardiovascular Surgery (PANDA IV)
Acronym: PANDA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Shanghai East Hospital of Tongji University (Other); West China Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Cardio-Thoracic Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PANDA IV
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease; Cardiopulmonary Bypass
Keywords: Gut microbiota
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fecal Microbiota Transplantation; Capsules

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of this research, we could not keep the participants blind to group assignment, but the study staff and statistical analyses were all blind to patient allocation during datacollection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intestinal Microbial Transformation (IMT) (Experimental): The Intestinal Microbial Transformation (IMT) group received Probacine, in addition to standard treatment and care, including prophylactic antibiotics , fluid therapy, and enteral nutrition supports.
  Interventions: Drug: Intestinal Microbiota Transplant (IMT) Capsules
- Control (No Intervention): The control group received standard treatment and care, including prophylactic antibiotics , fluid therapy, and enteral nutrition supports.

INTERVENTIONS:
Drug: Intestinal Microbiota Transplant (IMT) Capsules — Intestinal Microbiota Transplant (IMT) Capsules were administered 7 days preoperatively and 14 days postoperatively.
  Arms: Intestinal Microbial Transformation (IMT)

SUMMARY:
Cardiovascular diseases (CVDs) continue to be the primary cause of illness and death globally, emphasizing the pressing requirement for efficient prevention methods. Recent studies indicate that the gut microbiome plays a vital role in maintaining cardiovascular health, affecting the pathophysiological mechanisms related to CVDs. The potential therapeutic strategies for primary care practitioners included the modulation of the gut microbiome through dietary changes, prebiotics, and probiotics. The aim of this study was to investage the effect of gut microbiome modulation on clinical outcomes after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women;
* Cardiovascular surgery;
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Pregnant women;
* Patients with preexisting psychotic disorders;
* Decline to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Gastrointestinal Injury | 14 days after surgery

SECONDARY OUTCOMES:
ΔSOFA | 7 days after surgery
  the difference between the mean total postoperative SOFA score and baseline score within 24 hours of surgery during the index admission
30-day mortality rate | 30 days after surgery
  defined as mortality within 30 days postoperatively in the hospital or anywhere after discharge;

CONTACTS AND LOCATIONS:
Overall Officials: Guo-liang Fan, Study Director — Shanghai East Hospital
Locations (5):
- China (5):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Shanghai East Hospital, Tongji University, Shanghai

IPD SHARING:
Plan to Share IPD: No